Official Title: A Phase IIb, Randomized, Double-Blind, Placebo-Controlled,

Multicenter Study to Evaluate the Efficacy and Safety of Intravenous Prasinezumab in Participants with Early Parkinson's Disease

NCT Number: NCT04777331

**Document Date:** Statistical Analysis Plan Version 2: 05-Aug-2024

#### STATISTICAL ANALYSIS PLAN

STUDY TITLE: A PHASE IIB, RANDOMIZED, DOUBLE-BLIND,

PLACEBO-CONTROLLED, MULTICENTER STUDY TO EVALUATE THE EFFICACY AND SAFETY OF INTRAVENOUS PRASINEZUMAB IN PARTICIPANTS

WITH EARLY PARKINSON'S DISEASE

STUDY NUMBER: BN42358

STUDY NAME: PADOVA

VERSION NUMBER: 2

**ROCHE COMPOUND:** Prasinezumab (RO7046015)

**EUDRACT NUMBER:** 2020-004997-23

**IND NUMBER:** 119602

NCT NUMBER: NCT04777331

PLAN PREPARED BY: , PhD

#### STATISTICAL ANALYSIS PLAN APPROVAL

SPONSOR: F. Hoffmann-La Roche Ltd
LEGAL REGISTERED Grenzacherstrasse 124
ADDRESS: 4070 Basel, Switzerland

**DATE FINAL:** See electronic date stamp on the last page of this

document

#### **CONFIDENTIAL**

This is an F. Hoffmann-La Roche Ltd document that contains confidential information. Nothing herein is to be disclosed without written consent from F. Hoffmann-La Roche Ltd.

Prasinezumab—F. Hoffmann-La Roche Ltd Statistical Analysis Plan BN42358

# STATISTICAL ANALYSIS PLAN VERSION HISTORY

This statistical analysis plan (SAP) was developed based on Roche SAP model document Version (v)2.0.

| SAP Version | Approval Date | Based on Protocol<br>(Version, Approval Date) |
|---|---|---|
| 1 | 12 <sup>th</sup> April 2024 | v4.0, 30 October 2023 |
| 2 | see electronic date stamp<br>on the last page of this<br>document | v4.0, 30 October 2023 |

# STATISTICAL ANALYSIS PLAN AMENDMENT, VERSION 2: RATIONALE

<u>The SAP of BN42358 has been amended to incorporate the</u> FDA comments received in June 2024 on the SAP v1 submitted on the 19<sup>th</sup> of April 2024.

• Changes to the SAP, along with a rationale for each change, are summarized below: Section 4.6.4 from SAP version 1 was merged with Section 4.2.2. The new section has been renamed to change in symptomatic PD treatment.



# **TABLE OF CONTENTS**

| 1. | | INTRODUCTION | 10 |
|----|-------|------------------------------------------------------|----|
| | 1.1 | Objectives and Endpoints | 10 |
| | 1.2 | Study Design | 12 |
| | 1.2.1 | Treatment Assignment | 13 |
| | 1.2.2 | Blinding | 13 |
| | 1.2.3 | Data Monitoring | 14 |
| 2. | | STATISTICAL HYPOTHESES AND SAMPLE SIZE DETERMINATION | 14 |
| | 2.1 | Statistical Hypotheses | 14 |
| | 2.2 | Sample Size Determination | 14 |
| | 2.3 | Analysis Timing | 15 |
| 3. | | ANALYSIS SETS | 15 |
| 4. | | STATISTICAL ANALYSES | 16 |
| | 4.1 | General Considerations | 16 |
| | 4.1.1 | Definition of Baseline | 16 |
| | 4.2 | Primary Analysis | 16 |
| | 4.2.1 | MDS-UPDRS Definition | 16 |
| | 4.2.2 | Change in Symptomatic PD Treatment | 16 |
| | 4.2.3 | Primary Endpoint Analyses | 18 |
| | 4.2.4 | Main Analytical Approach for Primary Endpoint | 18 |
| | 4.2.5 | Stratification and Covariates for Adjustment | 19 |
| | | | 19 |
| | 4.2.7 | Sensitivity Analyses | 20 |
| | | | 20 |
| | | | 21 |
| | 4.3 | Statistical Analyses for Secondary Endpoints | 21 |
| | | | 22 |
| | | | 22 |
| | | | 23 |
| | 4.4 | Exploratory Efficacy Analyses | 23 |

| | 4.4.1 | Digital Biomarker Analysis Plan | <mark>25</mark> |
|---|---|---|---|
| | 4.4.2 | EQ-5D-5L | 25 |
| | 4.5 | Safety Analyses | 25 |
| | 4.5.1 | Extent of Exposure | 26 |
| | 4.5.2 | Adverse Events | 26 |
| | | | 26 |
| | 4.5.4 | Laboratory Data | 27 |
| | 4.5.5 | Vital Signs and ECG | 27 |
| | 4.6 | Other Analyses | 27 |
| | 4.6.1 | Summaries of Conduct of Study | 27 |
| | 4.6.2 | Summaries of Treatment Group Comparability/Demographics and Baseline Characteristics | 27 |
| | 4.6.3 | Previous and Concomitant Medications | 27 |
| | 4.6.4 | Pharmacokinetic Analyses | 28 |
| | 4.6.5 | Immunogenicity Analyses | 29 |
| | 4.6.6 | Biomarker Analyses | 29 |
| | | | 30 |
| | 4.8 | Interim Analyses | |
| | 4.9 | Changes to Protocol- planned Analyses | |
| 5. | | SUPPORTING DOCUMENTATION | |
| 6. | | REFERENCES | 33 |
| | | LIST OF TABLES | |
| <u>Ta</u> | ble 1 | Primary Objective and Estimand Definition | 10 |
| Ta | ble 3 | Participant Analysis Sets | |
| | | | 19<br>20 |

# **LIST OF FIGURES**

| Figure 1 | Study Schema. | 13 |
|----------|---------------|-----|
| | | 2 1 |

## LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

A2R adenosine receptor subtype 2

ADA anti-drug antibody

ADBL analysis database lock

AE adverse event

AESI adverse event of special interest

ANCOVA analysis of covariance

ATC anatomical therapeutic chemical

ATT Average Treatment Effect in the Treated

AUC area under curve

C-SSRS Columbia-Suicide Severity Rating Scale

CCOD clinical cutoff date

CGI-C Clinician Global Impression of Change

CGI-S Clinician Global Impression of Severity

CI confidence interval

C<sub>max</sub> maximum concentration

C<sub>trough</sub> trough concentration

COMT catechol-o-methyl-transferase

CSF cerebrospinal fluid

CSR Clinical Study Report

d-BAP digital Biomarker Analysis Plan

DAP Data Analysis Plan

DaT-SPECT dopamine transporter with single photon emission computed

tomography

ECG electrocardiogram

EQ-5D-5L EuroQoL 5-Dimension 5-Level questionnaire

FAS full analysis set

FDA U.S. Food and Drug Administration

H&Y Hoehn and Yahr

HR hazard ratio

IAS immunogenicity analysis set

iDMC independent Data Monitoring Committee

IMP investigational medicinal product

IRR infusion-related reaction

IV intravenous

IxRs interactive voice/web-based response system

L-Dopa levodopa

LEDD levodopa equivalent daily dose

LoPO list of planned outputs

MAO-B monoamine oxidase B

MAR missing at random

MDD minimum detectable difference

MDS-UPDRS Movement Disorder Society - Unified Parkinson's Disease Rating

Scale

MedDRA Medical Dictionary for Regulatory Activities

MIDD Model Informed Drug Development

MMRM mixed model for repeated measures



NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

NONMEM non-linear mixed effects modeling

OLE open-label extension

PAS pharmacokinetic analysis set

PD Parkinson's disease

PGI-C Patient Global Impression of Change

PGI-S Patient Global Impression of Severity

PK pharmacokinetic

PPMI Parkinson's progression markers initiative

PS propensity score

PSM patient symptom measure

PT preferred term

Q4W every 4 weeks

REM rapid eye movement

SAE serious adverse events

SAP Statistical Analysis Plan

SAS safety analysis set

SMD standardized mean differences

SOC System Organ Class

SSS simple sum score

SDTM Study Data Tabulation Model

SDTMv Study Data Tabulation Model view

TTE time to event

V version

WHO World Health Organization

# 1. INTRODUCTION

This Statistical Analysis Plan (SAP) covers the analyses planned for the randomized double-blind treatment period. Analyses will be listed directly in the corresponding list of planned outputs (LoPO). The description of layouts for the Clinical Study Report (CSR) outputs, the details about the underlying analysis datasets and programs, with the linking production outputs to sections in the CSR are not within the scope of this document and will be covered in separate documents, i.e., Data Analyses Plan (DAP) Modules 2 and 3. The analyses as part of the open-label extension (OLE) and the comparison of the OLE to an external comparator arm is also described in this updated version 2 of this SAP.

The analyses described in this SAP will further detail and supersede those specified in Protocol BN42358 (hereafter referred to as PADOVA) and will be reported in the primary CSR.

### 1.1 OBJECTIVES AND ENDPOINTS

Please see the study protocol (Section 2) for details on the study objectives and endpoints.

The Estimand definition for the primary objective is detailed in Table 1.

 Table 1
 Primary Objective and Estimand Definition

| Primary Objective | Estimand Definition |
|---|---|
| prasinezumab compared with placebo (in participants on stable symptomatic monotherapy with either MAO-B inhibitors or L-Dopa, irrespective of their increase in | Population: Participants with early PD on stable symptomatic monotherapy with either MAO-B inhibitors or L-Dopa. |
| | Endpoint: Time to a confirmed motor progression event from the randomization date. Confirmed motor progression is defined as the first time point of a worsening event, defined either by: |
| | <ul> <li>A≥5 points increase in MDS-UPDRS Part III<br/>score (assessed in "OFF" medication state)<br/>from baseline sustained over two consecutive<br/>assessments,</li> </ul> |
| | OR |
| | <ul> <li>LEDD increase (see Section 4.2.2), after the first occurrence of "a≥5-points increase in MDS-UPDRS Part III score (assessed in "OFF" medication state) from baseline, and before any subsequent MDS-UPDRS Part III assessment.</li> </ul> |
| | <u>Treatment:</u> |

| Primary Objective | Estimand Definition |
|---|---|
| | Experimental arm: prasinezumab, administered as a 1500 mg IV infusion Q4W (in addition to the symptomatic monotherapy). |
| | Control arm: placebo, administered as an IV infusion Q4W (in addition to the symptomatic monotherapy). |
| | Population-level summary: hazard ratio of a confirmed motor progression event in MDS-UPDRS Part III score ("OFF" medication state) comparing the prasinezumab arm vs placebo. |

IV = intravenous; L-Dopa=levodopa; LEDD = levodopa equivalent daily dose; MAO-B=monoamine oxidase B inhibitors; MDS-UPDRS = Movement Disorder Society-Unified Parkinson's Disease Rating Scale; PD=Parkinson's disease; Q4W = every 4 weeks.





The secondary exploratory as well as pharmacokinetic (PK), immunogenicity, biomarker and safety objectives and endpoints are summarized in the study protocol. Their statistical analyses are further detailed in Section 4.3, Section 4.4, Section 4.5 and Section 4.6.

#### 1.2 STUDY DESIGN

PADOVA, is a randomized, double-blind, placebo-controlled, parallel group, multicenter study to evaluate efficacy and safety of prasinezumab, administered as 1500 mg intravenous (IV) infusion every 4 weeks (Q4W), to participants with early Parkinson's disease (PD) on stable symptomatic monotherapy (monoamine oxidase B [MAO-B] inhibitor or levodopa [L-Dopa]). See Figure 1 (study schema) for description of the study periods.



Please refer to Protocol Section 3 for further details regarding the study design.

Figure 1 presents an overview of the study design.

Figure 1 Study Schema



OLE= open-label extension.

## 1.2.1 <u>Treatment Assignment</u>

This is a randomized, double-blind study. After initial written informed consent was obtained, all screening procedures and assessments completed, and eligibility established (see Protocol Sections 4.1.1 and 4.1.2) for a participant, the study site received the participant's identification number and treatment assignment from an interactive voice/web-based response system (IxRS).

Participants were randomly assigned to one of two treatment arms: prasinezumab or placebo with study drug administered Q4W. Randomization occurs in a ratio through use of a permuted-block randomization method to ensure a balanced assignment to each treatment arm. Randomization is stratified according to the following criterion: PD medication (MAO-B vs. L-Dopa).

## 1.2.2 Blinding

Once the double-blind treatment period of the study is completed, participants who consent and are eligible will enter the OLE portion of the trial and will receive prasinezumab for approximately 2 years. Participants and sites will remain blinded to prior randomization assignment until the end of the OLE period.

All participants will be asked to come back for a safety follow-up visit after the end of the double-blind treatment period (for participants not enrolling in the OLE), or at the end of the OLE (for participants enrolling in the OLE).

All participants who discontinue treatment or withdraw from the study early (during the double-blind treatment period) will be asked to return approximately 28 days ( $\pm 7$  days) after the final dose of study drug in order to complete the early termination visit.

In addition, participants who prematurely discontinue from the study treatment will be asked to return for collection of safety and efficacy data according to the schedule of activities until the end of the double-blind treatment period. These participants will also be asked to participate in end-of-study and safety follow-up visits.

After the end-of-study visit or early termination visit, adverse events (AEs) should be recorded as outlined in Protocol Sections 5.5 and 5.6.

Refer to the schedule of activities (see Appendix 1 in the Protocol) for the list of assessments to be performed at the safety follow-up visit.

## 1.2.3 <u>Data Monitoring</u>

This study utilizes an independent Data Monitoring Committee (iDMC) to evaluate participant safety. Relevant efficacy data may be reviewed by the iDMC as part of risk/benefit assessments. More details on the role and process of the iDMC can be found in the iDMC charter.

# 2. <u>STATISTICAL HYPOTHESES AND SAMPLE SIZE</u> <u>DETERMINATION</u>

## 2.1 STATISTICAL HYPOTHESES

The hypotheses to be tested for the primary estimand are:

| • |
|---|
| • |

The null hypothesis will be tested at (with the randomization stratification factor as defined in Section 4.2.5).

If the primary endpoint is met, the secondary endpoints will be tested confirmatory according to a (see Section 4.3).

## 2.2 SAMPLE SIZE DETERMINATION

The purpose of this study is to investigate the effect of prasinezumab on time to clinical disease progression, defined as a confirmed motor progression on Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III score (in "OFF" medication state for participants on L-Dopa background therapy).



A total of 575 participants were planned to be recruited into the study within 11 months and 586 participants were actually randomized in this study.

#### 2.3 ANALYSIS TIMING



# 3. ANALYSIS SETS

The analysis population for the efficacy analyses is the full analysis set (FAS) consisting of all randomized participants, with participants grouped according to their randomized treatment.

The safety analysis set (SAS) consists of all randomized participants who received at least one dose of study drug, with participants grouped according to treatment received.

The analysis population for the pharmacokinetic analysis set (PAS) consists of all randomized participants exposed to study treatment with sufficient dosing information and at least one adequately documented and quantifiable prasinezumab concentration.

The immunogenicity analysis set (IAS) consists of all participants on active treatment with at least one anti-drug antibody (ADA) assessment.

The participant analysis sets are summarized in Table 3.

**Table 3 Participant Analysis Sets** 

| Participant<br>Analysis Set | Description |
|---|---|
| FAS | All randomized participants according to the treatment they were randomized to. |
| SAS | All randomized participants exposed to study treatment according to the treatment received. Participants will be summarized in the active treatment arm if they received at least one dose of study drug. |
| PAS | All randomized participants exposed to study treatment with sufficient dosing information and at least one adequately documented and quantifiable prasinezumab concentration. |
| IAS | All participants on active treatment with at least one ADA assessment. |

ADA = anti-drug antibody; FAS = full analysis set; IAS = immunogenicity analysis set;

PAS = pharmacokinetic analysis set; SAS = safety analysis set.

## 4. STATISTICAL ANALYSES

## 4.1 GENERAL CONSIDERATIONS

All statistical tests will be conducted at a

# 4.1.1 <u>Definition of Baseline</u>

For all efficacy analyses (including summaries of demographic characteristics as well as change from baseline), baseline will be defined as the assessment taken at the randomization date.

For all safety analyses, the baseline will be defined as the last pre-dose assessment prior to the first drug intake. If this baseline assessment does not exist, an earlier assessment will be taken.

## 4.2 PRIMARY ANALYSIS

## 4.2.1 MDS-UPDRS Definition

The MDS-UPDRS is a multimodal scale consisting of four subscales (Parts I-IV), see Protocol Section 4.5.5.1.

## 4.2.2 Change in Symptomatic PD Treatment

It is expected that during the conduct of this trial, participants change their regimen of symptomatic PD treatment and it is considered as a concomitant event.

The dosage of all reported symptomatic PD treatments will be converted to a LEDD using the methods described in Tomlinson 2010 and Jost and Kaldenbach 2023.



# 4.2.3 <u>Primary Endpoint Analyses</u>

The primary efficacy endpoint is time to a confirmed motor progression, defined as:

 A 5-points increase in MDS-UPDRS Part III score (assessed in "OFF" medication state) from baseline sustained over two consecutive assessments (regardless of the amount of time in between these two consecutive assessments),

OR

• LEDD increase (see Section 4.2.2), after the occurrence of a 5-points increase in MDS-UPDRS Part III score (assessed in "OFF" medication state) from baseline, and before any subsequent MDS-UPDRS Part III assessment (the first LEDD increase from the day of the occurrence of a 5-points progression and prior to the next assessment is considered to complete the event definition).

, see

Section 4.2.6 for handling of the missing data.

Participants who had a confirmed motor progression event remain in the study and continue to receive double-blind study treatment without any changes in their schedule of assessments.

The population summary measure for the primary endpoint is the HR of a confirmed motor progression between prasinezumab and placebo as defined in Section 1.1 (see Table 1).

# 4.2.4 Main Analytical Approach for Primary Endpoint

Disease progression curves in each treatment arm will be estimated using Kaplan–Meier methodology. The treatment effect will be quantified via a HR, computed from a stratified Cox proportional-hazards regression model, including a 95% confidence interval (CI).

A check of the proportional hazards assumption will be performed by plotting the log negative log of the estimated survivor function against log time.

Sensitivity analyses for the primary endpoint are described in Section 4.2.7.

# 4.2.5 <u>Stratification and Covariates for Adjustment</u>

For the primary analyses a stratified log-rank test and stratified Cox proportional hazards model will be conducted. In addition, the following covariates will be used in a supplementary analysis for the primary endpoint, as well as for secondary and exploratory endpoint analyses, further specified in Section 4.3 and Section 4.4: 1. 2. 3. 4. 5.



# 4.2.7 <u>Sensitivity Analyses</u>

The following sensitivity analysis will be performed in the FAS:

• The primary analysis will be repeated using an unstratified log-rank test.





## 4.3 STATISTICAL ANALYSES FOR SECONDARY ENDPOINTS

If the primary endpoint is met, secondary endpoints

If the statistical significance of the primary endpoint is not reached, p-values will be interpreted descriptively.

The secondary endpoints will be tested in the FAS in the following confirmatory order provided the null hypothesis of the primary endpoint is rejected:

- 1. Change in motor function from baseline to Week 76, as measured by the MDS-UPDRS Part III score (assessed in "OFF" medication state).
- 2. Change in bradykinesia and rigidity from baseline to Week 76, as measured by the MDS-UPDRS Part III bradykinesia and rigidity, sum of the two subscores (assessed in "OFF" medication state).
- 3. Time to meaningful worsening (defined as a rating of "very much worse," "much worse," or "minimally worse") in Clinician Global Impression of Change (CGI-C, Overall Disease Subscale).
- 4. Time to onset (≥ 1 point increase from baseline) of motor complications as assessed through MDS-UPDRS Part IV.

- Time-to-worsening of participant's motor function as reported by the participant
  (≥ 3 points increase in MDS-UPDRS Part II score from baseline) in the presence of
  a confirmed motor progression event.
- 6. Time to meaningful worsening (defined as a rating of "very much worse," "much worse," or "minimally worse") in Patient Global Impression of Change (PGI-C, Overall Disease Subscale).



Missing scores for the corresponding endpoint will not be imputed; they will be handled via the MMRM model. The MMRM assumes that missing data are missing at random (MAR). That is, MMRM assumes that given the statistical model and given the observed values of the endpoint, the missing data are independent of the unobserved values (O'Kelly and Ratitch 2014). Correlation between successive observations on a subject allows data from subjects who dropped out to make a contribution to the estimation of the effects at the final time point.





# 4.4 EXPLORATORY EFFICACY ANALYSES

The following TTE exploratory endpoints will be analyzed for the FAS using the same statistical methodology as defined for the primary endpoint (Section 4.2):

The following change from baseline exploratory endpoints will be analyzed in the FAS using the same statistical methodology as defined for the secondary endpoints using MMRM (see Section 4.3):



The following additional endpoints will be analyzed in the FAS using a MMRM with the model specifications as described in Section 4.3:





4.4.1 Digital Biomarker Analysis Plan

The following exploratory endpoints will be analyzed:



A separate digital Biomarker Analysis Plan (d-BAP) will list and describe the motor and cognitive digital assessments performed using the Roche PD Mobile Application, v3.0, the single features to be extracted and analyzed, the patient-reported impression of motor symptom severity (smartphone PGI-S), along with the framework and methods used to build and analyze the simple sum score (SSS) and the patient symptom measure (PSM). The d-BAP will cover in detail the pre-processing steps that will be applied to digital sensor feature data, the analysis objectives, and the statistical methods used to analyze the single features, smartphone PGI-S and SSS.

The results from all the above-mentioned analyses will be reported separately and outside of the main study CSR.

### 4.4.2 EQ-5D-5L

The EuroQoL 5-Dimension 5-Level questionnaire (EQ-5D-5L) will be analyzed separately outside of SAP and will be reported outside of the CSR.

#### 4.5 SAFETY ANALYSES

Descriptive statistics (including percentages and frequencies for categorical data, means and medians, standard deviations for continuous data) using the SAS will be used to analyze the safety data collected in the double-blind treatment period (Table 3).

The following safety and tolerability analyses will be conducted:

- Nature, incidence, seriousness and severity of AEs, with severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
- Incidence of AEs of special interest.

- Incidence of treatment discontinuations due to AEs.
- Nature, incidence, seriousness, severity, and timing of infusion-related reactions (IRRs).
- Mean change in vital signs from baseline over time and incidence of abnormal vital sign measurements.
- Changes in electrocardiogram (ECG) assessments from baseline over time and incidence of abnormal ECG assessments.
- Change from baseline and incidence of laboratory abnormalities (including hematology, clinical chemistry, coagulation, and urinalysis parameters).
- Shift tables of laboratory abnormalities (including hematology, clinical chemistry, coagulation, and urinalysis parameters).
- Change from baseline in suicidal ideation, as measured by Columbia-Suicide Severity Rating Scale (C-SSRS).

## 4.5.1 Extent of Exposure

Exposure to prasinezumab and placebo over the course of the study will be summarized using descriptive statistics for the safety population by treatment as follows:

- Treatment duration (weeks).
- Total number of administrations.
- Total cumulative dose (mg).
- Number of doses.
- Planned dose.
- Missed doses (by AE/other).

## 4.5.2 <u>Adverse Events</u>

Verbatim descriptions of treatment-emergent AEs will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) in effect at the time of analysis database lock (ADBL). A treatment-emergent AE is defined as any new AE or any worsening of an existing condition with an onset date on or after the first study drug administration date.

Incidence in participant years and overview summaries of AEs, related AEs, serious adverse events (SAEs), AEs by greatest intensity/severity (NCI CTCAE) grade, AEs related to study drug, adverse event of special interest (AESI), ADA, risks and IRRs will be provided by System Organ Class (SOC) and preferred term (PT) where applicable.



## 4.5.4 Laboratory Data

Laboratory data will be summarized by treatment group for each assessment visit using descriptive statistics of absolute values, change from baseline values, and percentage change from baseline. In addition, incidence of laboratory abnormalities (including hematology, clinical chemistry, coagulation, and urinalysis parameters) will be summarized by treatment group, visit and baseline status. Shift tables for laboratory abnormalities will be provided.

## 4.5.5 Vital Signs and ECG

Absolute values and change from baseline values for vital signs and ECG will be summarized by descriptive statistics at each visit by treatment group. Incidence of abnormal vital signs and ECG measurements will be summarized descriptively by visit. Shift tables for vital signs and ECG will be provided too.

#### 4.6 OTHER ANALYSES

# 4.6.1 Summaries of Conduct of Study

The number of participants who enrolled, discontinued, or completed the study will be summarized by treatment arm. Reasons for premature study discontinuation will be listed and summarized. Enrollment, number of major protocol deviations (overall and by the standard four main categories: inclusion criteria, exclusion criteria, medication and procedural) and number of investigational medicinal product (IMP) administrations will be summarized by treatment arm. Participant disposition will be summarized by treatment arm and will include whether treatment was completed or discontinued early, and the reason for early treatment discontinuation.

# 4.6.2 <u>Summaries of Treatment Group Comparability/Demographics</u> <u>and Baseline Characteristics</u>

Demographic and baseline characteristics (including age, sex, symptomatic treatment, disease duration, number of years of education, race and/or ethnicity, and H&Y stage) will be summarized descriptively for the FAS (see Table 3).

Descriptive summaries of continuous data will present the means, standard deviations, medians, and minimum and maximum. Descriptive summaries of categorical data will include frequencies and percentages of participants.

# 4.6.3 <u>Previous and Concomitant Medications</u>

Previous medications recorded before screening until the start of treatment will be presented in summary tables as well as the concomitant medications.

The original terms recorded in the clinical database by the Investigator for concomitant medications will be standardized by the Sponsor using the WHO Drug dictionary.

## 4.6.4 Pharmacokinetic Analyses

Participants data (for the PAS, see Table 3) will be included in the PK analyses if there is sufficient dosing information and at least one adequately documented and quantifiable prasinezumab concentration per participant.

The population PK model (Report 1081130) initially developed with the Phase I data of prasinezumab and subsequently updated with PASADENA PK data, will be used to analyze the sparse sampling dose-concentration-time data of prasinezumab collected during this study. Non-linear mixed effects modeling (with software NONMEM [Beal and Sheiner 1998]) will be used. Structural model refinement will be driven by the data and will be based on various goodness of fit indicators. The model may be revised if necessary.

Population and individual PK parameters (e.g., clearance and central volume) will be estimated and the influence of different covariates

will be investigated. Secondary PK parameters such as area under curve (AUC), maximum concentration ( $C_{max}$ ) and trough concentration ( $C_{trough}$ )at steady state will be derived from the individual post-hoc predictions.

Additional PK analyses will be conducted as appropriate.

Graphical exploration of the relationship between prasinezumab exposure and disease progression (assessed by a confirmed motor progression) will be performed. If indicated by such exploration, more formal analyses of the PK/pharmacodynamic relationship using non-linear mixed effects modeling methods will be conducted.

Exploratory analyses will also be performed in order to explore:

- The relationship between serum concentration or secondary PK parameters of prasinezumab and other efficacy endpoints.
- The relationship between serum concentration or secondary PK parameters of prasinezumab and biomarker endpoints.
- The relationship between serum concentration or secondary PK parameters of prasinezumab and safety endpoints.



## 4.6.5 Immunogenicity Analyses

As ADA samples from participants assigned to the placebo group will not be analyzed for prasinezumab PK concentration in the first instance, except by request, only the treated group will undergo statistical analysis in the first instance. The immunogenicity analysis population will be conducted on IAS (see Table 3).

The numbers and proportions of ADA-positive participants and ADA-negative participants at baseline (baseline prevalence) and after drug administration (post-baseline incidence) will be summarized by treatment group. When determining post-baseline incidence, participants are considered to be ADA positive if they are ADA negative or have missing data at baseline but develop an ADA response following study drug exposure (treatment-induced ADA response), or if they are ADA positive at baseline and the titer of one or more post-baseline samples is at least 4-fold greater than the titer of the baseline sample (treatment-enhanced ADA response). Participants are considered to be ADA negative if they are ADA negative or have missing data at baseline and all post-baseline samples are negative, or if they are ADA positive at baseline but do not have any post-baseline samples with a titer that is at least 4-fold greater than the titer of the baseline sample (treatment unaffected).

The relationship between ADA status and safety, efficacy, PK, and biomarker endpoints may be analyzed and reported using descriptive statistics.

# 4.6.6 <u>Biomarker Analyses</u>

Based on FAS (depending on availability of biomarker assessment for individual participants), ANCOVA analyses (with covariates and stratification factor as defined in Section 4.2.5) are planned for the following:



Further exploratory biomarker analyses may be conducted separately (e.g. on ) for which separate analysis plans will be used.









#### 4.8 INTERIM ANALYSES

There is no plan to conduct any interim analysis.

## 4.9 CHANGES TO PROTOCOL- PLANNED ANALYSES

Not planned.

# 5. <u>SUPPORTING DOCUMENTATION</u>

This SAP is part of a broader DAP including DAP Module 2, and DAP Module 3. The LoPO will be described in the Roche DAP module 2.

## 6. REFERENCES

Beal SL, Sheiner LB. NONMEM users guide part VII: conditional estimation methods. NONMEM Project Group, 1998.

Buuren SV and Groothuis-Oudshoorn K. Mice: Multivariate Imputation by Chained Equations in R. Journal of Statistical Software, 2011; 45: 1-67.

Goetz CG, Luo S, Wang L, et al. Handling missing values in the MDS-UPDRS. Mov Disord. 2015 Oct; 30(12): 1632–1638.

Hirano, K., & Imbens, G. W. (2001). Estimation of causal effects using propensity score weighting: An application to data on right heart catheterization. Health Services and Outcomes Research Methodology, 2(3-4), 259-278.

ICH E9 (R1) addendum on estimands and sensitivity analysis in clinical trials to the guideline on statistical principles for clinical trials

ICH E9 statistical principles for clinical trials - Scientific guideline

Jost ST, Kaldenbach MA., Antonini A, et al Levodopa Dose Equivalency in Parkinson's Disease: Updated Systematic Review and Proposals. Movement Disorders, 2023; 38: 1236-52.

Lavielle M. Mixed Effects Models for the Population Approach: Models, Tasks, Methods and Tools (First edition). CRC Press, 2014.

Li, H., and Yue, L. Q. (2023). Propensity score-based methods for causal inference and external data leveraging in regulatory settings: From basic ideas to implementation. Pharmaceutical Statistics. https://doi.org/10.1002/pst.2294

Mallinckrodt, C.H., Bell, J., Liu, G. et al. Aligning Estimators With Estimands in Clinical Trials: Putting the ICH E9(R1) Guidelines Into Practice. Ther Innov Regul Sci 54, 353–364 (2020).

Marek K, Chowdhury S, Siderowf A, et al. Parkinson's Progression Markers Initiative. The Parkinson's progression markers initiative (PPMI) - establishing a PD biomarker cohort. Annals of Clinical and Translational Neurology, 2018; 5: 1460-77.

Marras C, Rochon P, Lang AE. Predicting Motor Decline and Disability in Parkinson Disease: A Systematic Review. Arch Neurol. 2002;59(11):1724–1728.

O'Kelly M, and Ratitch B. Clinical trials with missing data: a guide for practitioners. Chichester. John Wiley & Sons, 2014.

Pagano G, Taylor KI, Anzures Cabrera J, et al. Prasinezumab slows motor progression in rapidly progressing early-stage Parkinson's disease, Nature Medicine, 2024 Apr;30(4):1096-1103.

Poewe W, Seppi K, Tanner CM, et al. Parkinson disease. Nature Reviews Disease Primers, 2017; 3: 17013.

Politis M, Wu K, Molloy S, et al. Parkinson's disease symptoms: the patient's perspective. Movement Disorders, 2010; 15; 25(11): 1646-51.

Post B, Merkus MP, de Haan RJ, Speelman JD; CARPA Study Group. Prognostic factors for the progression of Parkinson's disease: a systematic review. Mov Disord. 2007 Oct 15;22(13):1839-51; quiz 1988.

Ratitch B. and O'Kelly M. Implementation of Pattern-Mixture Models Using Standard SAS/STAT Procedures. Proceedings of PharmaSUG, 2011.

Rosenbaum, PR., and Rubin, DB. "The Central Role of the Propensity Score in Observational Studies for Causal Effects." Biometrika, vol. 70, no. 1, 1983, pp. 41–55.

Spillantini MG, Schmidt ML, Lee VM, et al. Alphasynuclein in Lewy bodies. Nature, 1997; 388(6645): 839-40. doi:10.1038/42166. PMID: 9278044.

Sprenger F, Poewe W. Management of motor and non-motor symptoms in Parkinson's disease. CNS Drugs, 2013; 27: 259-72.

Stephenson D, et al. Transforming Drug Development for Neurological Disorders: Proceedings from a Multidisease Area Workshop. Neurotherapeutics, 2023; 20: 1682-91.

Thomas, L. E., Li, F., and Pencina, M. J. Overlap weighting: A propensity score method that mimics attributes of a randomized clinical trial. JAMA,2020; 323(23), 2417-2418. https://doi.org/10.1001/jama.2020.7819

Tomlinson CL, Stowe R, Patel S, et al. Systematic review of levodopa dose equivalency reporting in Parkinson's disease, Movement Disorders, 2010; 25(15): 2649-53.

Westfall PH and Krishen A. Optimally weighted, fixed sequence and gatekeeper multiple testing procedures. Journal of Statistical Planning and Inference, 2001; 99: 25–40.

1081130. Population pharmacokinetic and pharmacokinetic-pharmacodynamic analyses of RO7046015 in healthy subjects (Study PRX002-CL001) and Parkinson's Disease patients (Study PRX002-CL002). August 2017.

# Signature Page for Statistical Analysis Plan - BN42358 - Published System identifier: RIM-CLIN-617627

| Approval Task | |
|---------------|-------------------------------|
| | Company Signatory |
| | 05-Aug-2024 07:09:05 GMT+0000 |